CLINICAL TRIAL: NCT06905587
Title: Effect of Methylphenidate on Cancer-related Fatigue in Patients Treated for a Brain Tumor During Childhood or Adolescence: Protocol for a Randomized, Double-blind, Placebo-controlled Crossover Trial - the EMBRAIN Trial
Brief Title: Methylphenidate in Pediatric Brain Tumor Survivors With Cancer-related Fatigue
Acronym: EMBRAIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Aalborg University Hospital (Other); Rigshospitalet, Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24/51848; R352-A20781 (Other Grant/Funding Number: The Danish Cancer Society); 2023-001094 (Other Grant/Funding Number: The Danish Childhood Cancer Foundation); 2023-507926-18-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-27; First posted 2025-04-01 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor, Pediatric; Cancer-related Fatigue; Methylphenidate
Keywords: methylphenidate; cancer-related fatigue; brain tumor; childhood cancer; pediatric cancer; childhood cancer survivor; late effect; long-term effects secondary to cancer therapy in children; long-term effects of cancer-treatment; pediatric brain tumor
MeSH Terms: conditions — Brain Neoplasms; Neoplasms | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylphenidate, Then Placebo (Experimental): Patients will receive treatment with methylphenidate tablets for 6 weeks, and then cross over to treatment with methylphenidate-matched placebo tablets for an additional 6 weeks. A four week wash out period is incorporated between treatments.
  Interventions: Drug: Methylphenidate (MPH); Drug: Placebo
- Placebo, Then Methylphenidate (Experimental): Patients will receive treatment with methylphenidate-matched placebo tablets for 6 weeks, and then cross over to treatment with methylphenidate tablets for an additional 6 weeks. A four week wash out period is incorporated between treatments.
  Interventions: Drug: Methylphenidate (MPH); Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate (MPH) — 10 mg methylphenidate tablets with a scoreline. Tablets will be administered orally.
  For children aged 6-12, a daily dose of 5 mg x 2 will be administered during the first week with an increase in dose to 10 mg x 2 in the second week. For adolescents and adults above 12 years of age, the same starting dose will be used as for children, with weekly incremental increases up to a maximum of 15 mg x 2 daily in the third week. In case of potential toxicity events during study, dosage of methylphenidate can be modified according to protocol.
Drug: Placebo — 10 mg methylphenidate-matched placebo tablets with a scoreline. Tablets will be administered orally.
  Dosage will follow the exact same principles as for the study drug (methylphenidate).

SUMMARY:
Cancer-related fatigue is a common and debilitating late effect in pediatric brain tumor survivors. Currently, evidence-based recommendations to ameliorate this condition are lacking.

The researchers will investigate the ability of methylphenidate to improve fatigue and cognition in pediatric brain tumor survivors suffering from cancer-related fatigue. Methylphenidate is a drug (central nervous stimulant) most commonly used in the treatment of hyperkinetic disorders such as attention-deficit/hyperactivity disorder (ADHD).

If methylphenidate shows an effect, the prospects are important for this patient group, since methylphenidate may then be included as part of the treatment of brain tumor-related fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed and treated for a brain tumor during childhood or adolescence (0-≤18 years).
2. Treated for a PBT during the previous 10 years, starting from date of diagnosis.
3. Aged ≥6 years 0 months at the start of the trial.
4. Off therapy/active treatment for pediatric brain tumor (PBT) for 12 months at the start of the trial.
5. No known signs of clinical or radiological tumor progression at last follow-up.
6. Danish is the sole or primary language (enabling provision of validated assessment tools).
7. Patient and family have provided consent for inclusion in the trial.
8. Clinically significant fatigue based on the PedsQL MFS questionnaire at baseline, defined by a score ≥ 1 standard deviation below the normative mean.
9. History of clinically relevant fatigue after treatment of PBT compared to estimated premorbid ability, as assessed from consultations in the childhood cancer outpatient clinics.

Exclusion Criteria:

1. Any known contraindications to methylphenidate as outlined below:

   A) Hypersensitivity to the active substance or any excipients listed in the summary of product characteristics. B) Glaucoma. C) Pheochromocytoma. D) Hyperthyroidism. E) Mania. F) Psychosis. G) Anorexia nervosa. H) Current or previous severe depression. I) Suicidal behavior. J) Poorly controlled type 1 bipolar affective disorder. K) Antisocial or borderline personality disorder. L) Pre-existing cardiovascular disorders, including severe hypertension, heart failure, arterial occlusive disease, angina pectoris, hemodynamically significant congenital heart disease, cardiomyopathies, myocardial infarction, potentially life-threatening cardiac arrhythmias and channelopathies. M) Pre-existing cerebrovascular disease, cerebral aneurysm, vascular abnormalities including vasculitis or stroke. N) Treatment with irreversible MAO inhibitors within the last 14 days and reversible MAO inhibitors within the last 24 hours.
2. History of recent poorly controlled seizures.
3. Motor tics or Tourette syndrome (including family history of tic disorder).
4. Known diagnosis of Attention Deficit/Hyperactivity Disorder or Autism Spectrum Disorder.
5. Known diagnosis of Full Scale Intelligence Quotient (FSIQ) of <50.
6. Pregnancy. Participants known to be pregnant or breastfeeding at screening/registration will not be enrolled in the trial. All sexually active women of childbearing potential (WOCBP) must have a negative pregnancy test prior to the start of treatment. Acceptableeffective contraceptive must be used for the duration of the trial. No further testing is needed during trial, unless the participant suspects to have become pregnant.
7. Concerns about family ability to safely store or administer MPH, or to report side effects appropriately/concerns about familial substance abuse.
8. Concurrent use of opiods (ATC N02A) or benzodiazepines (ATC N05BA and N05CF).
9. Simultaneously enrolled in another clinical trial investigating cancer-related fatigue with a pharmaceutical intervention.

Ages: 6 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
PedsQL Multidimensional Fatigue Scale (MFS) | At baseline, at Week 6, Week 16, and Week 20 (follow-up).
  Changes in patient self-reported fatigue (participants above 18 years of age) or parent proxy-reported fatigue (participants between 6-17 years of age) from baseline to week 6 of MPH or placebo treatment as measured by the PedsQL Multidimensional Fatigue Scale (MFS).

SECONDARY OUTCOMES:
PedsQL Multidimensional Fatigue Scale (MFS) | At baseline, at Week 6, Week 16, and Week 20 (follow-up).
  Changes from baseline in self-reported fatigue (participants aged 6-17 years of age) measured by the PedsQL MFS.
Behaviour Rating Inventory of Executive Function (BRIEF) | At baseline, at Week 6, and Week 16.
  Changes from baseline in self and parent-reported executive function measured by the BRIEF-2 or BRIEF-V questionnaire.
Connor's Continuous Performance Test (CPT) Online Suite | At baseline, at Week 6, and Week 16.
  Changes from baseline in digital measures of sustained attention and executive function. CPT-3 and K-CPT-2 will be used.
Wechsler Coding | At baseline, at Week 6, and Week 16.
  Changes from baseline in processing speed. Coding module from Wechsler Intelligence Scale for Children Fifth Edition (WISC-V) or Wechsler Adult Intelligence Scale Fifth Edition (WAIS-V) depending on age of participant.
Wechsler Digit Span | At baseline, at Week 6, and Week 16.
  Changes from baseline in working memory. Coding module from WISC-V or WAIS-V depending on age of participant.
PedsQL Generic Core Scales | At baseline, at Week 6, and Week 16.
  Changes from baseline in self and parent-reported measures of Health Related Quality of Life.
Accelerometry (Axivity AX3) | Accelerometry will be performed for a duration of 1 week during week 4-6 and week 14-16 during the study arm.
  Time spent within different activity domains and sleep-wake patterns measured by accelerometry. Axivity AX3 accelerometers will be used.
Barkley's Stimulant Side Effect Rating Scale (SSERS) | At baseline, Week 2, Week 3, Week 4, Week 6, Week 10, Week 12, Week 13, Week 14, Week 16, and Week 20 (follow-up)..
  Changes from baseline in self and parent-reported side-effects. A modified version of SSERS with 21 items customized to Danish practice will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Rathe, Consultant, MD, PhD, Study Director — Odense University Hospital
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No